CLINICAL TRIAL: NCT05058183
Title: Safe De-escalation of Chemotherapy for Stage 1 Breast Cancer
Acronym: Safe-De
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Massachusetts General Hospital (Other); Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCR5348
Record Dates: First submitted 2021-08-19; First posted 2021-09-27 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is looking into the ctDNA diagnostic test, this is given after breast cancer surgery to see whether patient is clear from cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants
  Interventions: Diagnostic Test: ctDNA

INTERVENTIONS:
Diagnostic Test: ctDNA — Patients with stage 1 HER2 positive and triple negative breast cancer will receive ctDNA test after surgery. Treating clinicians will receive results and may change treatment plans in event of negative test.

SUMMARY:
The aim of this study is to assess the rates of circulating tumour DNA (ctDNA) in patients treated with surgery for stage 1 breast cancer that is HER2 positive or triple negative.

The study will involve collecting blood samples from patients before and after surgery, if patients are enrolled after surgery, blood samples will be collected after the procedure. On the follow-up visit, the results obtained from the blood tests will serve as a diagnostic method to discern adverse outcomes in the groups of patients with positive and negative ctDNA detection. Also, the results obtained will aid physicians in determining treatment courses for patients, in order to reduce the intensity of adjuvant chemotherapy. By identifying the patients with residual disease with ctDNA analysis, it is possible that this will improve disease prognosis.

DETAILED DESCRIPTION:
Patients with stage 1 breast cancers have a very good prognosis, with the substantial majority cured by local therapy alone. However, the vast majority of HER2 positive and triple negative breast cancers (TNBC) with stage 1 (T1b and T1c) disease receive adjuvant chemotherapy after surgery. To reduce morbidity shorter courses of chemotherapy have become the standard. For HER2 positive breast cancer twelve weeks of weekly taxol and trastuzumab has very good long term outcomes, with only 1% of patients having a distant recurrence at seven year follow-up. Similarly for triple negative breast cancer four cycles of chemotherapy, for example with the docetaxel-cyclophosphamide regimen, may be used. This compares to the use of full adjuvant chemotherapy for HER2 positive breast cancer for example 4 cycles of anthracycline-cyclophosphamide chemotherapy followed twelve weeks of weekly taxol with trastuzumab and pertuzumab, and full (neo)adjuvant chemotherapy for TNBC of 4 cycles of anthracycline-cyclophosphamide chemotherapy followed twelve weeks of weekly taxol with carboplatin.

Detection of circulating tumour DNA (ctDNA) in plasma, after treatment for primary breast cancer, is associated with a very high risk of future relapse. As cancer cells proliferate and die, a small amount of cancer cell DNA is released into blood circulation. Sequencing of the primary cancer to identify the mutations present in the cancer, allows very sensitive detection of these mutations in DNA extracted from plasma. Detection of cancer specific mutations in the plasma DNA implies that there is cancer present in the body. For patients who have already had potentially curative treatment for breast cancer, detection of cancer specific mutations or ctDNA, identifies the presence of molecular residual disease, and that this residual disease is proliferating. The identification of ctDNA in these patients is associated with a very high risk of future relapse.

As most patients with stage I breast cancer are cured by the surgery alone, it is not possible on a population basis to discern adverse outcomes with reducing the intensity of adjuvant chemotherapy, by offering shorter courses of chemotherapy. Yet for those few patients who will relapse without chemotherapy, those with molecular residual disease, short-course chemotherapy increases their risk of relapse compared to full combination adjuvant chemotherapy. Yet in routine clinical practice there is no way of identifying who has molecular residual disease. If we can identify who the patients with residual disease with ctDNA analysis, those patients can escalate treatment to full chemotherapy and thereby improve their outcome.

The Signatera assay identifies the presence of molecular residual disease with high accuracy in many tumour types. Patients with ctDNA detected have a very high risk of future relapse. The assay is available as a routine validated clinical test, of proven clinical validity. The purpose of this study is to allow patients to access the Signatera assay as part of their standard clinical care, and to identify which patients have a high risk of relapse after treatment for stage I breast cancer by detecting the presence of ctDNA after surgery, who would have a higher risk of relapse if treated with short-course chemotherapy.

Patients will be enrolled into the study prior to surgery, in preference, to shorten the time from surgery to the ctDNA testing result being available. Patients will also have a ctDNA test taken prior to surgery, to explore whether this result may also have prognostic significance. The pre-surgery result will not be made available to patients or their treating clinicians in this study, as the full clinical importance of this result is not as clear as detection after surgery.

This protocol describes a study that will be conducted in the United Kingdom, and a parallel protocol will recruit patients in the United States sponsored by Massachusetts General Hospital. The two protocols share the same objectives and statistical design and endpoints, although are tailored to the individual health care systems. The sample size describes the combined recruitment of the protocols, and the databases of the two protocols will be combined for assessment of all endpoints. The study will aim to recruit a minimum of 40% of patients from each country (up to 200 patients from each country).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Patients with histologically confirmed breast cancer that is either

   A) HER2 positive as defined by 2018 ASCO-CAP guidelines determined by local testing B) Triple negative defined as ER negative (ER staining in <1% tumour cells or ER Allred score <3/8) and PR negative (PR staining in <10% tumour cells or PR Allred score <6/8) and HER2 negative by 2018 ASCO-CAP guidelines determined by local testing. Patients without PR testing results may enrol on the basis of ER and HER2 results.

   Note that patients negative for ER and PR may enrol whilst awaiting HER2 testing results
3. Stage 1 cancer excluding pT1aN0 cancer, defined as

   A) Patients prior to surgery with primary tumour size on imaging 6-20mm and a normal axilla ultrasound or a biopsy negative axilla

   Patients who enrol prior to surgery will only continue further testing in the trial if their pathological staging fits the after surgery criteria.

   B) Patients after surgery with either
   * Primary tumour size pT1b or pT1c (6-20mm) and pN0 or pN1mi (micrometastasis).
   * Primary tumour size pT1a (1-5mm) and pN1mi

   Note that patients consenting after surgery may not enrol with pT1aN0 stage disease
4. Patients should consent prior to surgery (preferred) or within 2 weeks of surgery. Patients who consent after surgery may extend consent to 4 weeks after surgery, although this will delay the receipt of ctDNA results.
5. Planned and fit enough to receive full standard post-operative chemotherapy, with HER2 targeting as appropriate.
6. Ability to give informed consent and comply with study procedures including blood tests and follow-up for five years.

Exclusion Criteria:

1. Distant metastatic disease.
2. Multifocal invasive cancer
3. Diagnosis of alternative cancer within the last 5 years other than resected non-melanoma skin cancer or cervical intraepithelial neoplasia.
4. Any prior treatment (including neo-adjuvant chemotherapy) for the current breast cancer with the exception of surgical resection for patients enrolling after surgery.
5. Known HIV or hepatitis B or hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2028-12-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients with ctDNA detection treated with surgery for stage 1 breast cancer | 2 to 4 weeks post surgery.
  Blood samples will be analysed for the presence of circulating tumour DNA using the standard clinical Signatera assay.

SECONDARY OUTCOMES:
Relapse free survival | Through study completion, minimum 5 years unless early study termination.
  The time from the date of surgery to relapse in the ipsilateral breast, nodal regions, or with distant metastatic disease, or death from any cause. Disease free patients and second cancers will be censored at study closure date.
Proportion of physicians who change treatment advice | Up to 6 weeks post surgery.
  Determined by questionnaire responses.
Distant recurrence free survival | Through study completion, minimum 5 years unless early study termination.
  The time from the date of surgery to relapse with distant metastatic disease or death from any cause. Local recurrence and second cancers would be censored.
Invasive disease free survival | Through study completion, minimum 5 years unless early study termination.
  The time from the date of surgery to local or distant breast cancer invasive recurrence, new breast cancer ipsilateral or contralateral, or death from any cause. Non-invasive recurrences and second cancers would be censored.
Overall survival | Through study completion, minimum 5 years unless early study termination.
  Time from randomisation to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Turner, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, Chelsea, London
  - The Royal Marsden NHS Foundation Trust, Sutton, Sutton

REFERENCES:
- [Background] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Background] Coombes RC, Page K, Salari R, Hastings RK, Armstrong A, Ahmed S, Ali S, Cleator S, Kenny L, Stebbing J, Rutherford M, Sethi H, Boydell A, Swenerton R, Fernandez-Garcia D, Gleason KLT, Goddard K, Guttery DS, Assaf ZJ, Wu HT, Natarajan P, Moore DA, Primrose L, Dashner S, Tin AS, Balcioglu M, Srinivasan R, Shchegrova SV, Olson A, Hafez D, Billings P, Aleshin A, Rehman F, Toghill BJ, Hills A, Louie MC, Lin CJ, Zimmermann BG, Shaw JA. Personalized Detection of Circulating Tumor DNA Antedates Breast Cancer Metastatic Recurrence. Clin Cancer Res. 2019 Jul 15;25(14):4255-4263. doi: 10.1158/1078-0432.CCR-18-3663. Epub 2019 Apr 16. PMID 30992300
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Garcia-Murillas I, Chopra N, Comino-Mendez I, Beaney M, Tovey H, Cutts RJ, Swift C, Kriplani D, Afentakis M, Hrebien S, Walsh-Crestani G, Barry P, Johnston SRD, Ring A, Bliss J, Russell S, Evans A, Skene A, Wheatley D, Dowsett M, Smith IE, Turner NC. Assessment of Molecular Relapse Detection in Early-Stage Breast Cancer. JAMA Oncol. 2019 Oct 1;5(10):1473-1478. doi: 10.1001/jamaoncol.2019.1838. PMID 31369045
- [Background] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Background] Jones S, Holmes FA, O'Shaughnessy J, Blum JL, Vukelja SJ, McIntyre KJ, Pippen JE, Bordelon JH, Kirby RL, Sandbach J, Hyman WJ, Richards DA, Mennel RG, Boehm KA, Meyer WG, Asmar L, Mackey D, Riedel S, Muss H, Savin MA. Docetaxel With Cyclophosphamide Is Associated With an Overall Survival Benefit Compared With Doxorubicin and Cyclophosphamide: 7-Year Follow-Up of US Oncology Research Trial 9735. J Clin Oncol. 2009 Mar 10;27(8):1177-83. doi: 10.1200/JCO.2008.18.4028. Epub 2009 Feb 9. PMID 19204201
- [Background] Loibl S, O'Shaughnessy J, Untch M, Sikov WM, Rugo HS, McKee MD, Huober J, Golshan M, von Minckwitz G, Maag D, Sullivan D, Wolmark N, McIntyre K, Ponce Lorenzo JJ, Metzger Filho O, Rastogi P, Symmans WF, Liu X, Geyer CE Jr. Addition of the PARP inhibitor veliparib plus carboplatin or carboplatin alone to standard neoadjuvant chemotherapy in triple-negative breast cancer (BrighTNess): a randomised, phase 3 trial. Lancet Oncol. 2018 Apr;19(4):497-509. doi: 10.1016/S1470-2045(18)30111-6. Epub 2018 Feb 28. PMID 29501363
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Background] Tolaney SM, Barry WT, Dang CT, Yardley DA, Moy B, Marcom PK, Albain KS, Rugo HS, Ellis M, Shapira I, Wolff AC, Carey LA, Overmoyer BA, Partridge AH, Guo H, Hudis CA, Krop IE, Burstein HJ, Winer EP. Adjuvant paclitaxel and trastuzumab for node-negative, HER2-positive breast cancer. N Engl J Med. 2015 Jan 8;372(2):134-41. doi: 10.1056/NEJMoa1406281. PMID 25564897
- [Background] Tolaney SM, Guo H, Pernas S, Barry WT, Dillon DA, Ritterhouse L, Schneider BP, Shen F, Fuhrman K, Baltay M, Dang CT, Yardley DA, Moy B, Marcom PK, Albain KS, Rugo HS, Ellis MJ, Shapira I, Wolff AC, Carey LA, Overmoyer B, Partridge AH, Hudis CA, Krop IE, Burstein HJ, Winer EP. Seven-Year Follow-Up Analysis of Adjuvant Paclitaxel and Trastuzumab Trial for Node-Negative, Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer. J Clin Oncol. 2019 Aug 1;37(22):1868-1875. doi: 10.1200/JCO.19.00066. Epub 2019 Apr 2. PMID 30939096
- [Background] von Minckwitz G, Procter M, de Azambuja E, Zardavas D, Benyunes M, Viale G, Suter T, Arahmani A, Rouchet N, Clark E, Knott A, Lang I, Levy C, Yardley DA, Bines J, Gelber RD, Piccart M, Baselga J; APHINITY Steering Committee and Investigators. Adjuvant Pertuzumab and Trastuzumab in Early HER2-Positive Breast Cancer. N Engl J Med. 2017 Jul 13;377(2):122-131. doi: 10.1056/NEJMoa1703643. Epub 2017 Jun 5. PMID 28581356